CLINICAL TRIAL: NCT05363696
Title: Paulista Cardiovascular Surgery Registry (REPLICCAR)
Brief Title: The REPLICCAR Registry and The Statewide Quality Improvement Initiative
Acronym: REPLICCAR
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto do Coração do Hospital das Clinicas da Faculdade de Medicina da Universidade de São Paulo (Unknown); Hospital Samaritano Paulista (Other); Hospital Israelita Albert Einstein (Other); Beneficência Portuguesa de São Paulo (Other); Instituto Dante Pazzanese de Cardiologia (Other); Hospital das Clinicas da Universidade Estadual de Campinas (Unknown); Hospital de Base de São Jose do Rio Preto (Unknown); Irmandade da Santa Casa de Misericórdia de Marília (Unknown); Irmandade da Santa Casa de Misericórdia de São Paulo (Unknown); Irmandade da Santa Casa de Misericórdia de Piracicaba (Unknown); Hospital São Paulo da Universidade Federal de São Paulo (Unknown); Hospital Pitangueiras do Grupo SOBAM (Unknown); Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - USP (Unknown)
Responsible Party: Sponsor
Other Study IDs: 450617006
Record Dates: First submitted 2022-05-02; First posted 2022-05-06 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2019-05

CONDITIONS: Cardiac Surgical Procedures
Keywords: Database; Quality improvement; Mortality; Coronary artery bypass grafting; Heart valve surgery
MeSH Terms: interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Coronary artery bypass grafting (CABG) — Coronary artery bypass grafting surgery procedure
Procedure: Heart valve surgery — Heart valve surgery procedure

SUMMARY:
Cardiovascular diseases remain the leading cause of death for the healthcare system and cardiac surgery has an important impact on their resolubility. Healthcare systems in the world have evolved to optimize their clinical records and thus learn from the real world through the interactivity between results, processes, and structure. When the rate of growth of healthcare costs scenario is greater than the one of Gross Domestic Product of countries, there is a considerable challenge to increment the quality of healthcare services and the primordial patient safety, as well as the necessary control and traceability of implantable devices. The association and correlation of patients' demographic and clinically relevant information with the resources required for the care provided for each stratum represent the possibility to adapt, improve and innovate the healthcare programs; This will allow improving the optimization of the therapeutic protocols and the creation of related research areas, aiming to promote more equitable resources allocation, increase access and effectiveness, as well as to ascertain the magnitude of available and used resources and its impact.

DETAILED DESCRIPTION:
METHODS Extension Cohort study, mandatory, prospective multicenter, in the state of São Paulo and of registry of consecutive cases. Besides the situational diagnostic of the results and comparison between the mean of both registries, there will be the creation of improvement reports for each of the REPLICCAR centers.

Next, quality improvement initiatives will be implemented in each center indicated by the reports.

Sample

* Will be included in a consecutive way all patients that had CABG and heart valve surgery in the participant centers for the defined period;
* Data will be collected, independently of surgical volume, severity status, and social condition among others, in sight of the São Paulo state health department;
* This way, it will be possible to produce a predictive curve to be used in most clinical case scenarios observed in the state of São Paulo;

ELIGIBILITY:
Inclusion Criteria:

* Age 18- 90 years old.
* CABG or heart valve surgery
* Agreement to participate in the study signing informed consent documentation.

Exclusion Criteria:

* Re-operation
* Impossibility to access data variables relevant to the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18-90 years old) underwent cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 9723 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Create and implementing data driven quality initiatives for cardiac surgery procedures in São Paulo state | 5 years
  Guided by the database, quality initiatives will be built in order to reduce mortality, length of stay and complications in the centers participating in REPLICCAR.

SECONDARY OUTCOMES:
Create a morbidity and mortality risk score | 5 years
  Create a morbidity and mortality risk score, in order to guide the care and interventions of patients undergoing cardiac procedures, in order to prevent morbidity and mortality outcomes.
Long-term follow-up of patients included in the database | 10 years
  Long-term follow-up of patients included in the database, providing an opportunity to assess quality of life, evolution and deaths after hospital discharge.
Assessment of the impact of patients' socioeconomic variation in its surgical evolution | 10 years
  Assessment of the impact of patients' socioeconomic variation on their evolution in terms of morbidity and mortality (short and long term).

CONTACTS AND LOCATIONS:
Overall Officials: Omar AV Mejia, MD,PhD, Principal Investigator — USP Heart Institute
Locations (2):
- Brazil (2):
  - USP Heart Institute, São Paulo
  - Fabio B Jatene, MD, PhD, São Paulo

IPD SHARING:
Plan to Share IPD: No
The Comissão de Ética para Análise de Projetos de Pesquisa (CAPPesq) - HC-FMUSP https://www.hc.fm.usp.br/index.php?option=com_content&view=article&id=243:comissao-de-etica-para-analise-de-projetos-de-pesquisa-do-hcfmusp&catid=23&Itemid=229 ) approved this analysis as part of the Project: "Surgical Risk Stratification as an Instrument for Innovation in Cardiac Surgery Programs in the Unified Health System of the São Paulo State " (REPLICCAR 1) under online registration Nº.450617006. This retrospective analysis was performed without identifying the patients. Therefore, patients' informed consent form was waived.

REFERENCES:
- [Result] Orlandi BMM, Mejia OAV, Borgomoni GB, Goncharov M, Rocha KN, Bassolli L, Melo de Barros E Silva PG, Nakazone MA, Sousa A, Campagnucci VP, de Sousa Vilarinho KA, Katz M, Tiveron MG, Arrais Dos Santos M, Lisboa LAF, Dallan LAO, Jatene FB; REPLICCAR II Study Group. REPLICCAR II Study: Data quality audit in the Paulista Cardiovascular Surgery Registry. PLoS One. 2020 Jul 10;15(7):e0223343. doi: 10.1371/journal.pone.0223343. eCollection 2020. PMID 32649718
- [Derived] Borgomoni GB, Dias RD, de Barros E Silva PGM, Nakazone MA, de Oliveira MAP, Campagnucci VP, Tiveron MG, Lisboa LAF, Hajjar LA, Zubelli JP, Jatene FB, Mejia OAV; REPLICCAR study group. Incidence of failure-to-rescue after coronary artery bypass grafting: a multicenter observational study from the REPLICCAR II registry in Brazil. Patient Saf Surg. 2025 Feb 11;19(1):6. doi: 10.1186/s13037-024-00417-9. PMID 39934891